CLINICAL TRIAL: NCT05352347
Title: A Randomized, Double-blinded, Placebo-controlled, Parallel-treatment Group, Adaptive Design, Multi-center, Phase 2b/3 Trial to Evaluate Efficacy and Safety of NuSepin® Intravenous Infusion in COVID-19 Pneumonia Patients
Brief Title: Phase 2b/3 Trial of NuSepin® in COVID-19 Pneumonia Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaperon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShaperonC002
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NuSepin® 0.2 mg/kg (Active Comparator): NuSepin® 0.2 mg/kg in 100mL NS bid
  Interventions: Drug: NuSepin® 0.2 mg/kg
- NuSepin® 0.4 mg/kg (Active Comparator): NuSepin® 0.4 mg/kg in 100mL NS bid
  Interventions: Drug: NuSepin® 0.4 mg/kg
- Placebo (Placebo Comparator): Normal saline (NS) 100mL bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NuSepin® 0.2 mg/kg — NuSepin® 0.2 mg/kg in 100mL NS bid
  Arms: NuSepin® 0.2 mg/kg
Drug: NuSepin® 0.4 mg/kg — NuSepin® 0.4 mg/kg in 100mL NS bid
  Arms: NuSepin® 0.4 mg/kg
Drug: Placebo — Normal saline (NS) 100mL bid
  Arms: Placebo

SUMMARY:
A Randomized, Double-blinded, Placebo-controlled, Parallel-treatment Group, Adaptive Design, Multi-center, Phase 2b/3 Trial to Evaluate Efficacy and Safety of NuSepin® Intravenous Infusion in COVID-19 Pneumonia Patients

ELIGIBILITY:
Inclusion Criteria:

1. An individual who or whose legally authorized representative has fully informed of all pertinent aspect of the trial and IMP, voluntarily decided to participate in the trial and adherence to the trial-related requirements, and provided a written informed consent
2. An adult man or woman aged between 19 years (or age of majority in his/her country) and 80 years.
3. A hospitalized patient with laboratory-confirmed SARS-CoV-2 infection by PCR test within 10 days (240 hours) prior to randomization.
4. At the time of randomization; whose clinical status is stage 4 (oxygenation by facial mask or nasal cannula) or 5 (non-invasive ventilation or high flow oxygen) on WHO 8-point ordinal scale
5. Pneumonia that satisfies all the following criteria at the time of randomization
6. Planned first dosing of the IMP not later than 2 days after the initiation of standard of care (SOC), when given in combination with SOC for severe Illness (according to NIH Clinical Spectrum of SARS-CoV-2 Infection)
7. A score of 5 points or more ("think sepsis") on the NEWS 2 scale at the time of randomization

Exclusion Criteria:

1. A patient whose clinical status is stage 3 or lower on the WHO 8-point ordinal scale (WHO 8-OS) at the time of randomization
2. An individual who requires endotracheal intubation, mechanical ventilation (WHO 8-OS stage 6), or extracorporeal membrane oxygen therapy (stage 7) at the time of randomization
3. A patient with multiorgan failure, shock, acute respiratory syndrome (ARDS)
4. A patient with renal dysfunction defined by eGFR less than 30mL/min/1.73m², or the use of hemodialysis or hemofiltration
5. Cholestatic liver disease (example: biliary obstruction, cholangitis, etc.) or hepatic dysfunction
6. Any of the following laboratory test results at the time of screening:
7. An individual with HIV-positive results or who requires antiviral treatments against active hepatitis (HBV, HCV) and etc.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to improvement of at least 2 categories relative to the first dosing date of the Investigational Medicinal Product (randomization date) on an 8-point ordinal scale (WHO 8-point ordinal scale) of clinical status up to day 29 [Phase 2b] | Day 29
Time to discharge relative to the first dosing date of the IMP (randomization date) [Phase 3] | Day 29

SECONDARY OUTCOMES:
WHO 8-point ordinal scale | Day 29
  The proportion of subjects with categories of 2 or less (outpatient condition); and 3 or less (hospitalized, no oxygen treatment) at day 8, 15 and 29 and etc.
NEWS 2 | Day 29
  Time to normalization of vital signs that lasts 24 hours or more (score 0 on NEWS2 that lasts 24 hours or more) and etc.
the use of ventilatory assistance | Day 29
  The proportion of subjects undergoing a ventilatory assistance (facial mask, low-flow oxygen cannula, high-flow oxygen cannula, Non-invasive ventilation, Invasive Mechanical Ventilation/ECMO) at day 8, day 15, and day 29; and the days of each ventilatory assistance since the first dosing date of IMP (randomization date) up to day 29
Hospitalization and ICU Admission | Day 29
  Proportion of subjects transferred to ICU and the duration of ICU admission (date of admission to ICU ~ discharge date) since the first dosing date of IMP (randomization date) up to day 29 and etc.
Survival | Day 29
  All-cause mortality; follow-up until discharge, or up to 60 days for patients who are still hospitalized at day 29 of the first IMP dosing (randomization date)
biomarkers | Day 29
  Proportions of subjects whose inflammatory-related biomarkers at baseline, day 4, day 8, day 15, day 29 are within the normal range (① TNF-α, ② IL-1β, ③ IL-6, ④ IL-8 ⑤ IL-18 ⑥ CRP) and etc.
Cytokine release syndrome | Day 29
  The proportion of subjects with a decrease of at least 1 category according to an ASTCT Consensus Grading step for Cytokine Release Syndrome
Viral burden | Day 29
  Proportion of patients who become negative for viral titer at each assessment time point since the first dosing date of IMP and etc.
Compliance | Day 29
  Compliance of the study drugs (days of dosing with the study drugs and total dose administered)
Safety Endpoints | Day 29
  The incidence and characteristics of adverse events after administration of IMP and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yong Seong, Dr., Study Chair — Shaperon Inc.
Locations (1):
- Gachon University Gil Medical Center, Incheon, Namdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No